CLINICAL TRIAL: NCT04111731
Title: Left Atrial Arrhythmia Substrate Identification by Ultra-high Density Mapping After Confirmed durABLE Pulmonary Vein Isolation
Brief Title: Left Atrial Arrhythmia Substrate Identification After Confirmed durABLE Pulmonary Vein Isolation
Acronym: LAUDABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200
Record Dates: First submitted 2019-04-03; First posted 2019-10-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: Radiofrequency catheter ablation; Cryoballoon pulmonary vein isolation; Rhythmia; Orion catheter; Posterior wall isolation; Electrophysiological study; Omron device
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A randomised, controlled multi-centre pilot study. Forty participants with persistent atrial fibrillation will have an equal chance of being randomised to receive either of two treatment techniques of pulmonary vein isolation:
  Cryoballoon (Group 1) or Radiofrequency ablation (Group 2). Subsequently, all patients will undergo a repeat procedure 2 months later to assess for reconnections requiring further treatment.
  In Group 2 participants, there will also be lesions made to the back wall of the heart (left atrial posterior wall isolation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group one (Active Comparator): Cryoballoon pulmonary vein isolation
  Interventions: Procedure: Cryoballoon pulmonary vein isolation; Procedure: Repeat electrophysiological study
- Group two (Active Comparator): Radiofrequency pulmonary vein isolation
  Interventions: Procedure: Radiofrequency pulmonary vein isolation; Procedure: Repeat electrophysiological study; Procedure: Left atrial posterior wall isolation

INTERVENTIONS:
Procedure: Cryoballoon pulmonary vein isolation — Catheter ablation using cryoballoon pulmonary vein isolation. Utilisation of a 'cold balloon' (Cryoenergy or cryoballoon ablation) to freeze the bases of the 4 pulmonary veins to achieve electrical isolation.
  Arms: Group one
Procedure: Radiofrequency pulmonary vein isolation — Catheter ablation using radiofrequency energy to achieve pulmonary vein isolation. Radiofrequency energy is delivered through the tip of a catheter to make tiny burns (ablation lesions) around the outlines of the 4 pulmonary veins at their bases
  Arms: Group two
Procedure: Repeat electrophysiological study — All participants will receive a repeat electrophysiological study 2 months after the index procedure during which radiofrequency catheter ablation guided by ultra-high density mapping will be used to identify regions of reconnection that need re-isolation; other tests will be carried out including testing for arrhythmia inducibility
  Other Names: Repeat catheter ablation
Procedure: Left atrial posterior wall isolation — The left atrial posterior wall will be isolated in Group 2 participants (those who received radiofrequency ablation at the index procedure) during the repeat electrophysiological study in 2 months
  Other Names: Posterior wall isolation
  Arms: Group two

SUMMARY:
Under current practice, patients with persistent atrial fibrillation, can be offered one of two types of ablation treatment. Both of these treatments are aimed at electrically isolating the 4 pulmonary veins (PVs) at the back of the heart which connect it to the lungs. These PVs have been identified to serve as the sites where the abnormal heart rhythm is generated. One of the treatments is called radiofrequency (RF) catheter ablation, where 'heat energy' is delivered through the tip of a catheter to make tiny burns (ablation lesions) around the outlines of the 4 PVs at their bases. The other treatment technique utilises a 'cold balloon' (Cryoenergy or cryoballoon ablation) to freeze the bases of the 4 PVs to achieve the electrical isolation. Sometimes the treated tissues develop reconnections that can lead to a recurrence of the abnormal heart rhythm, and thus the need for a repeat procedure.

In this study, participants will receive a second treatment 2 months after the first one. During the second treatment, investigators will check to identify areas that have developed reconnections since the first treatment; these will be treated again. This will increase the chances of all participants having a complete treatment.

In order to improve understanding of how best to treat this condition, investigators will also carry out some further measurements within the heart during the repeat procedure. During these measurements, investigators will check to see if treatment has succeeded in reducing the occurrence of an abnormal heart rhythm. In the group of participants in whom RF energy is used for the initial procedure, investigators will also treat the back wall of the heart, and repeat these measurements.

DETAILED DESCRIPTION:
Persistent atrial fibrillation (PeAF) is defined as continuous atrial fibrillation for 7 days or more. Approximately 10% of people are diagnosed with atrial fibrillation (AF) by age 80 years; and among people of European descent, 26% of men and 23% of women have a lifetime risk of developing AF after age 40.

Catheter ablation by pulmonary vein isolation is the usual approach employed for PeAF. This involves making lesions within the pulmonary veins to achieve electrical isolation. Electrical isolation cuts off abnormal electrical triggers originating from the pulmonary veins. However, treatment outcomes are less than optimal with a lot of variability in success rates for different techniques. Hence, the optimal treatment strategy for patients with PeAF is not clear.

In this pilot study, investigators aim to study two different treatment modalities of catheter ablation: cold balloon (cryoballoon, Group 1) and hot tip (radiofrequency ablation, Group 2) used in (electrically) isolating the pulmonary veins. There will be 1:1 randomisation to either of the two modalities. All participants will subsequently undergo a repeat procedure 2 months later to identify reconnections and to re-isolate the veins using the hot tip (radiofrequency ablation) guided by an ultra-high density mapping technology. During the repeat procedure, investigators will perform further electrophysiological studies including assessing arrhythmia inducibility and measuring the extent of isolated areas. For participants in Group 2, investigators will also make some lesions in the back wall of the heart (posterior wall isolation) and recheck arrhythmia inducibility.

All participants will be given a handheld ECG recording (Omron) device. Participants will be shown how to use the device to make daily 30-second recordings and when they have symptoms, to be reviewed. Follow up will be at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80 years
2. Evidence of persistent Atrial Fibrillation

Exclusion Criteria:

1. Any previous catheter (or surgical) ablation for atrial fibrillation or cryoballoon pulmonary vein isolation
2. An indwelling atrial septal defect (ASD) occluder device or anatomical structure that pre-vents free access to the left atrium
3. Left atrial diameter on transthoracic echo (Parasternal long axis, M-mode) > 5.5cm
4. Recent stroke/Transient Ischaemic Attack within 3 months
5. Inability, unwillingness or absolute contraindication to taking oral anticoagulant medication
6. Severe kidney impairment (estimated Glomerular Filtration Rate < 30ml/min)
7. Morbid obesity (Body Mass Index ≥40)
8. Extreme frailty
9. Severe valvular heart disease of any kind as assessed by the investigator, with or without prosthetic valve in place
10. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Number of late pulmonary vein re-connections | Up to 2 months after index ablation procedure
  Number of late pulmonary vein re-connections at repeat electrophysiological study as identified by ultra-high density mapping: comparison between the 80 pulmonary veins in each group

SECONDARY OUTCOMES:
Amount of radiofrequency energy needed to re-isolate the veins | 2 months after the index ablation procedure
  Amount of radiofrequency energy needed at repeat electrophysiological study to re-isolate the pulmonary veins
Area of low voltage | 2 months after the index ablation procedure
  Area of left atrial low voltage at start of repeat electrophysiological study under ultra-high density mapping guidance in each group
Incidence of arrhythmia inducibility before and after left atrial posterior wall isolation | 2 months after the index ablation procedure
  Incidence of arrhythmia inducibility after complete posterior wall isolation as compared to after pulmonary vein isolation alone assessed during an electrophysiological study
Incidence of peri-procedural complications | From index procedure to after repeat procedure
  Incidence of peri-procedural complications such as tamponade, major bleeding, myocardial infarction, requirement for permanent pacemaker, stroke, death
Incidence of renal function impacting on left atrial electrical properties | At the index procedure and 2 months after the index procedure
  Incidence of renal function impacting on electrical properties of the left atrium and arrhythmic substrate: assessed at baseline and during repeat electrophysiological study
Total length of time free from atrial arrhythmia estimated with the Omron device | At the 12th month follow-up visit
  Freedom from atrial arrhythmia at 12 months following the 2 procedures: comparison between groups. Time period free from atrial arrhythmia in minutes/hours/days
Quality of life assessment: validated questionnaire | At the index procedure and at the 6th month and 12th month follow-up appointments
  At baseline, 6 months and at 12 months using a validated questionnaire with 2 components: descriptive system and visual analogue scale. Descriptive system has 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each has 5 levels: no problems (level 1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5). The digits for the 5 dimensions will be combined into a 5-digit number describing the participant's health state - a total of 3125 possible health states. The health state will be converted to a single index value using conversion tables, and summarised as means or medians. Visual analogue scale records the participant's self-rated health on a 20 cm vertical scale with endpoints 'the best health you can imagine' and 'the worst health you can imagine'. It will be summarised as means or medians.
Clot formation and fibrinolysis assessment using turbidimetric analyses | At baseline, 2 months and 12 months
  Clot formation (lag time, rate of clot formation, maximum absorbance) and rate of fibrinolysis
Fibrin permeation testing | At baseline, 2 months and 12 months
  Permeation constant (Ks)

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MBBS MD FRCP, Study Chair — Liverpool Heart and Chest Hospital
Locations (3):
- United Kingdom (3):
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Manchester University NHS Foundation Trust, Manchester
  - The Newcastle Upon Tyne Hospital NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No